CLINICAL TRIAL: NCT04928014
Title: Validation of a Tear-based Screening Assay for Breast Cancer as a Supplemental Tool to Screening Mammograms
Brief Title: Validation of a Tear-based Screening Assay for Breast Cancer
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Namida Lab (Industry)
Responsible Party: Sponsor
Other Study IDs: Namida_001; PRO00053749 (Other: Advarra IRB)
Record Dates: First submitted 2021-06-09; First posted 2021-06-16 (Actual); Last update posted 2023-07-03 (Actual); Status verified 2023-06

CONDITIONS: Healthy; Breast Cancer; Breast Cancer Female; Health Care Utilization; Health Knowledge, Attitudes, Practice; Health Personnel Attitude; Health Care Acceptability
Keywords: preventative screening; protein biomarkers; lacrimal tear fluid; mammography; primary care; ELISA assay; CLIA laboratory; lab developed test; clinical utility; high complexity; underserved populations; health disparities; tear collection; mammogram; improved patient outcomes; reduces gap in access; health equity; total cost of care; trust from patient; increased compliance; affordable; non-invasive; women's health and wellness; breast health; breast cancer screening test
MeSH Terms: conditions — Breast Neoplasms; Patient Acceptance of Health Care; Behavior

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Lacrimal (tear) fluid
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Screening Mammogram: Individuals eligible for a screening mammogram.
  Interventions: Other: Schirmer Strip

INTERVENTIONS:
Other: Schirmer Strip — A tear-based screening assay for breast cancer developed and validated by Namida Lab, Inc., a high complexity CLIA-certified lab. It consists of two parts: tear sample collection using a Schirmer Strip and a clinical lab-developed test that measures protein biomarkers for breast cancer screening.

SUMMARY:
This study will explore and better understand the value, usage, and benefits of a tear-based screening test for breast cancer as a supplemental tool for screening mammograms. This tear-based screening test was developed and validated by Namida Lab, Inc., a high complexity Clinical Laboratory Improvement Amendments (CLIA) certified lab.

DETAILED DESCRIPTION:
The primary objective of this study is to determine if a tear-based biological test is an effective option in breast cancer screening. This will be assessed by comparing the score and classification produced from the assay to the current gold standard, screening Mammograms.

The primary endpoint will be assessed by calculating the sensitivity, specificity, PPV, and NPV for the biological assay compared to the results of imaging.

The secondary objective of this study is to obtain provider insight and recommendation as to the potential clinical utility of a tear-based biological test as a breast cancer screening option.

The secondary endpoint will be achieved through a provider roundtable discussion. After completion of enrollment and evaluation of tear samples and time will be arranged, either in person or virtual, to review the test scores determined for the sites patient population. Providers will be allowed to verbally review the process and give their thoughts on the utility of a tear-based biological test within their clinic and how they feel it should be used. A member of the Namida Lab clinical team will be present to take notes. After the discussion a report will be generated and the site providers will be allowed to review it for accuracy. Sites will be given a copy of their participants' scores as well as a summary of the provider roundtable discussion. Sites may request to have the participants' results blinded if prior to review if preferred.

ELIGIBILITY:
Inclusion Criteria:

Female over the age of 18 Able to undergo the informed consent process Willingness to comply with all study procedures

Exclusion Criteria:

Currently diagnosed or are receiving treatment for breast cancer Have an active eye infection under 18 years of age

Ages: 18 Years to 100 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Born biologically female
Study Population: The study population will be primarily women over the age of 35 who participate in yearly screening mammography. There are instances where a screening mammogram is given under the age of 35, therefore the enrollment age has been set at 18 years of age or older. Participants will be recruited from participating clinical sites which would include breast radiology speciality clinics, OB/GYN practice, internal medicine clinics, and primary care clinics.
Sampling Method: Non-Probability Sample
Enrollment: 205 (Estimated)
Dates: Start 2021-06-01 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Validation of a tear-based biological test | 3 years
  The primary endpoint will be assessed by calculating the sensitivity, specificity, PPV, and NPV for the a tear-based biological test compared to results of imaging

SECONDARY OUTCOMES:
Defining clinical utility of a tear-based biological test | 3 years
  The secondary objective of this study is to obtain provider insight and recommendation as to the potential clinical utility of a tear-based biological test as a breast cancer screening option.

CONTACTS AND LOCATIONS:
Locations (1):
- Namida Lab, Fayetteville, Arkansas, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Informed Consent Form (2021-05-10): https://cdn.clinicaltrials.gov/large-docs/14/NCT04928014/Prot_ICF_000.pdf